CLINICAL TRIAL: NCT02038192
Title: Living With Hope: Pilot Study of the Living With Hope Program for Family Caregivers of Persons With Dementia Residing in Long Term Care Facilities
Brief Title: Pilot Study of the Living With Hope Program for Family Caregivers of Persons With Dementia Residing in Long Term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00041954
Record Dates: First submitted 2013-10-04; First posted 2014-01-16 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Dementia
Keywords: Caregiver; Dementia; Long Term Care; Hope; Quality of Life; Intervention
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Living with Hope Program (Experimental): All participants in this group will receive the Living with Hope Program. It consists of viewing a 15 minute film on hope. Then for 5 minutes at the end of each day to write "Stories of the Present"to work on over one month. Stories of the present is a directed journaling activity which includes writing challenges of the day, what was their hope that day and what would be their hope tomorrow.
  Interventions: Behavioral: Living with Hope Program
- Stories of the Present (Experimental): Participants in this group will write Stories of the Present and not see the film.
  Interventions: Behavioral: Stories of the Present
- Usual Care (No Intervention): Participants in this group will not receive an intervention. Data collection for outcome variables will be the same as the participants in the other arms.

INTERVENTIONS:
Behavioral: Living with Hope Program — The Living with Hope Program is based on the research team's grounded theory study "Hope and Connection". The film " Connecting with Hope" reflects the findings of the grounded theory study. Stories of the Present has been utilized in the team's previous research with family caregivers of persons with advanced cancer.
  Arms: Living with Hope Program
Behavioral: Stories of the Present — Stories of the Present is a directed journaling activity in which participants write in a journal at the end of the day their challenges, hope and hope for tomorrow
  Arms: Stories of the Present

SUMMARY:
Hope is important for family/friends of persons with dementia residing in Long Term Care Facilities. Our research team has developed a program (Living with Hope) to increase hope and quality of life of family caregivers. The Living with Hope Program involves a) viewing the Living with Hope film which features caregivers of persons with dementia describing their hope and b) a hope activity entitled "Stories of the Present". A new Living with Hope film entitled "Connecting with Hope" has been produced and will be used in this pilot study. The purpose of this pilot study is to evaluate the feasibility and acceptability of the Living With Hope Program and collect preliminary data on the effectiveness of the Living with Hope Program for family members of persons with dementia residing in Long Term Care.

30 participants will be recruited from St. Joseph's Auxiliary hospital, the Alzheimer's Society of Alberta, and the Alberta Caregivers Association in Edmonton based on inclusion criteria. Participants will be randomly assigned to one of three groups: treatment (Watching a film on hope and Stories of the Present for one month); low dose group (Stories of the Present only); or usual care group. In all groups measures of hope, quality of life, self-efficacy and guild will be collected at visit 1, day 7, day 14 and one month in addition to demographic information. Participants in group 1 and 2 (treatment group) will be asked to describe what they were thinking about when doing the hope activities on day 7, 14 and one month using qualitative interviews. At one month all participants will be interviewed using open ended audio-taped questions to help evaluate the study procedures

DETAILED DESCRIPTION:
Background: Hope is important for family/friends of persons with dementia residing in Long Term Care Facilities (LTC). Our research team has developed a program (Living with Hope) to increase hope and quality of life of family caregivers. The Living with Hope Program (LWHP) involves a) viewing the Living with Hope film which features caregivers of persons with dementia describing their hope and b) a hope activity entitled "Stories of the Present". The hope activity consists of participants writing at the end of the day about their thoughts, challenges and what gave them hope over a 4- week time period. For family caregivers of persons with advanced cancer, this LWHP has been found to increase their hope and feelings of self-efficacy (confidence in their ability to deal with difficult situations). Based on a qualitative study of hope of family caregivers of persons with dementia residing in LTC, the LWHP has been adapted to that population. A new Living with Hope film entitled "Connecting with Hope" has been produced and will be used in this pilot study.

Aims: The purpose of this pilot study is to evaluate the feasibility and acceptability of the LWHP and collect preliminary data on the effectiveness of the Living with Hope Program for family members of persons with dementia residing in LTC.

Sample: Shannon Stachnik (Social Worker St. Joseph's Auxiliary Hospital), Arlene Huhn (Alzheimer's Society of Alberta - Edmonton) and Anna Mann (Alberta Caregivers Association) will identify potential participants based on the inclusion criteria. They will make contact and ask if the potential participants are willing to talk with a research nurse about the study. If they agree the research nurse will contact potential participants. Inclusion criterion for participants are: a) 18 years of age and older, b) English speaking, and c) have a family member or friend with dementia who resides in LTC.

The research nurse will contact potential participants and ask them when it will be a convenient time to meet with and obtain written informed consent.

Design: Using a mixed-methods randomized control trial (Quantitative +qualitative) design, 30 participants will be randomly assigned to one of three groups: 1) treatment (Watching a film on hope and Stories of the Present for one month), 2) low dose group (Stories of the Present only) or 3) usual care group. In all groups, demographic information, and baseline, day 7 ,14 and one month, measures of hope (Herth Hope Index), quality of life (WHOQOL-BREF), general self-efficacy (General Self-Efficacy Scale) and guilt (Caregiver Guilt Questionnaire) will be collected by a trained research nurse. Participants in group 1 and 2 (treatment group) will be asked to describe what they were thinking about when doing the hope activities on day 7, 14 and one month using qualitative interviews. At one month all participants will be interviewed using open ended audiotaped questions to help evaluate the study procedures

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* English speaking
* Have a family member or friend with dementia who resides in Long Term Care.

Exclusion Criteria:

* persons who are non-autonomous adults
* cognitively impaired as determined by the Registered Nurse (RN) researcher
* unable to participate, in the opinion of the RN researcher
* non-English speaking
* does not have a family member or friend with dementia in Long Term Care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hope | Change from baseline at day 7, 14 and 28
  Hope is measured by the Herth Hope Index (HHI). The Herth Hope Index is a 12 item (1-4 point)Likert scale that delineates three sub-scales of hope: a) temporality and future, b) positive readiness and expectancy, and c) interconnectedness. The HHI has been found to take approximately 5 minutes to complete. Summative scores range from 12-48, with a higher score denoting greater hope. The HHI has been found to be reliable (test-retest r=91, p<0.05) and valid (concurrent validity, r=84, p.,0.05; criterion, r=92, p,0.05; divergent, r=-0.73, p,0.05).

SECONDARY OUTCOMES:
Quality of Life | Change from baseline at day 7, 14 and 28
  Quality of Life is measured by the World Health Organization Quality of Life -Bref measure. The WHOQOL-BREF is a quality of life assessment measure based on the World Health Organization definition of quality of life reflecting 4 domains of quality of life: physical health (Domain 1), psychological health (Domain 2), social relations (Domain 3), and environment (Domain 4). The WHOQOL-BREF is comprised of 26 items measuring the domains and is a shorter version of the original WHOQOL. The scores are not reported as a total, but per domain. The higher the score, the higher the subjects' reported quality of life in each domain. Reliability has been reported to be 0.82. Cronbach's alpha for this scale was r = 0.76.

OTHER OUTCOMES:
General Self-efficacy | Change from baseline at day 7, 14 and 28
  General Self-efficacy is measured using the General Self-Efficacy Scale (GSES). This 10 item (0-4) Likert type scale produces a total perceived self-efficacy score. Higher scores on the GSES indicate a higher self-efficacy or the confidence of one's ability to deal with adverse situations. It has a maximum score of 40.
Caregiver guilt | change from baseline at day 7 , 14 and 28
  Caregiver guilt is measured by the Caregiver Guilt Questionnaire. This 22 item scale measures guilt on a five-point Likert scale (0 "Never" to 4 "Always") with a total range between 0 and 88. A higher score indicates that the respondent experienced more feelings of guilt related to their care giving. Cronbach's alpha indicated excellent internal consistency at 0.926.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy D. Duggleby, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada